CLINICAL TRIAL: NCT05760651
Title: Assessing Osteoporosis Awareness and Knowledge Levels In Turkish Multiple Sclerosis Patients: An Observational Study
Brief Title: Awareness of Osteoporosis in Multiple Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: OPMS1
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis; Osteoporosis; Osteoporosis Risk
MeSH Terms: conditions — Multiple Sclerosis; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis Patients: Patients diagnosed with multiple sclerosis.
  Interventions: Other: Patient Participation Form; Diagnostic Test: Timed up - and - go test

INTERVENTIONS:
Other: Patient Participation Form — A form that consists of revised osteoporosis knowledge test and osteoporosis awareness scale
Diagnostic Test: Timed up - and - go test — . The timed up-and-go test involves rising from a seated position, walking a distance of 3 meters, pivoting, returning to the initial point, and resuming a sitting position. It demonstrates strong inter-rater and intra-rater reliability, offering a reliable means of quantifying functional mobility and balance.

SUMMARY:
Osteoporosis is a condition that describes compromised skeletal microarchitecture in general, with clinical signs of decreased bone mineral density. Multiple sclerosis patients are at increased risk for developing osteoporosis. Identifying whether multiple sclerosis patients have information and awareness about this disease is crucial. This study is aimed to investigate awareness and knowledge of osteoporosis in multiple sclerosis (MS) patients. The study also aimed to assess potential differences and correlations in osteoporosis knowledge and awareness among MS patients based on gender, education levels, and risk of falls

DETAILED DESCRIPTION:
Osteoporosis is a common disease of bone loss. The reduced bone strength predisposes an increased risk for fractures in older individuals. It can affect people from different ethnicity. Many factors increase the risk of osteoporosis, including age, postmenopausal state, glucocorticoid use, low body weight, calcium, vitamin D, immobility, and chronic inflammation. Patients with multiple sclerosis are at high risk of developing osteoporosis due to chronic inflammation and their medications. Patients' knowledge and awareness about osteoporosis are essential for early detection, implementation of lifestyle changes, and treatment compliance. This study aimed to investigate osteoporosis awareness and knowledge about osteoporosis in patients with multiple sclerosis.The study also aimed to assess potential differences and correlations in osteoporosis knowledge and awareness among MS patients based on gender, education levels, and risk of falls

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of multiple sclerosis
* Must be between the ages of 18 and 99
* Must give consent to participate in the study

Exclusion Criteria:

• Not giving consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 90 years with a diagnosis of multiple sclerosis who gave consent to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Revised Osteoporosis Knowledge Test Scores | 1 day
  The 32-item Revised Osteoporosis Knowledge Test (ROKT; 2012), as reported by Gendler et al. (2015), is a revision of the original 24-item OKT developed by Kim, Horan, & Gendler (1991). This measure was developed to assess the osteoporosis knowledge of adults. Changes were made to update the original OKT to include current recommendations for calcium and vitamin D, exercise requirements, diagnosis and treatment, and a more comprehensive understanding of bone development and osteoporosis risk factors. It contains two subscales (Nutrition and Exercise), which share 14 common items including risk factors and general knowledge. Although the responses offered to participants are multiple choice (e.g., for risk items: more likely, less likely, neutral, don't know), there is only one correct answer for each item. Responses are dichotomously recoded as correct or incorrect.
Osteoporosis Awareness Scale Scores | 1 day
  The OAS, developed by Choi et al. in 2008, includes 31 items across 5 sub-dimensions, rated on a 4-point Likert scale. Validity and reliability assessment in Turkish was made by Aktürk et al. . The potential scores on the OAS range from a minimum of 31 to a maximum of 124. The overall osteoporosis awareness level is reflected in the mean score obtained from the entire scale, with higher scores indicating greater awareness. It's worth noting that the OAS doesn't include items with reverse scoring, and it lacks a specific cut-off point for interpretation.

SECONDARY OUTCOMES:
Correlation between the level of knowledge and awareness regarding osteoporosis with gender, education levels, and fall risks | 1 day
  Possible correlation will be analyzed using spearmans corelation test.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital
Locations (1):
- Sancaktepe Şehit Doktor İlhan Varank Training and Research Hospital, Istanbul, Sancaktepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon reasonable request.

REFERENCES:
- [Derived] Temel MH, Tasdelen B, Demir S, Ata E. Assessing osteoporosis awareness and knowledge levels of Turkish multiple sclerosis patients: an observational study. Arch Osteoporos. 2024 Aug 1;19(1):67. doi: 10.1007/s11657-024-01426-y. PMID 39085698